CLINICAL TRIAL: NCT06896916
Title: Phase 1/2 Study of Etentamig in Combination With a CELMoD Agent for the Treatment of Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Intravenously (IV) Infused Etentamig in Combination With an Oral Cereblon E3 Ligase Modulatory Drug (CELMoD) Agent Assessing Adverse Events and Change in Disease Activity in Adult Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-555; 2024-512146-41-00 (Other: EU CT)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cereblon E3 Ligase Modulatory Drug; CELMoD; Iberdomide; Etentamig; ABBV-383
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 1: ABBV-383 Dose Escalation (Experimental): In phase 1 participants will receive escalating Etentamig in combination with iberdomide, as part of the approximately 129 month study duration.
  Interventions: Drug: Etentamig; Drug: Iberdomide
- Phase 2: ABBV-383 Dose Expansion Dose A (Experimental): In phase 2 participants will receive Etentamig at dose A in combination with iberdomide, as part of the approximately 129 month study duration.
  Interventions: Drug: Etentamig; Drug: Iberdomide
- Phase 2: ABBV-383 Dose Expansion Dose B (Experimental): In phase 2 participants will receive Etentamig at dose B in combination with iberdomide, as part of the approximately 129 month study duration.
  Interventions: Drug: Etentamig; Drug: Iberdomide

INTERVENTIONS:
Drug: Etentamig — Intravenous (IV) Infusion
Drug: Iberdomide — Oral Capsule

SUMMARY:
Multiple myeloma (MM) is a plasma cell disease characterized by the growth of clonal plasma cells in the bone marrow. The purpose of this study is to assess the adverse events and change in disease activity of etentamig in combination with a cereblon E3 ligase modulatory drug (CELMoD) agent in adult participants with relapsed/refractory (R/R) multiple myeloma (MM). Adverse events and change in disease state will be assessed.

Etentamig is an investigational drug being developed for the treatment of R/R MM. Study doctors put the participants in groups called treatment arms. Multiple doses of etentamig in combination with iberdomide will be explored. Each treatment arm receives a different dose of etentamig and iberdomide to determine a tolerable dose. Approximately 135 adult participants with R/R MM will be enrolled in the study in approximately 50 sites worldwide.

In phase 1 participants will receive escalating intravenous (IV) etentamig in combination with oral iberdomide. In phase 2 participants will receive IV etentamig at one of two doses in combination with oral iberdomide, as part of the approximately 129 month study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and and monitoring of side effects.

DETAILED DESCRIPTION:
B-cell maturation antigen (BCMA) chimeric antigen receptor T-cell (CAR-T) or BCMA antibody-drug conjugate (ADC) are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance of 0 or 1.
* Must have confirmed diagnosis of Relapsed/Refractory Multiple Myeloma (RRMM) after the participant's last treatment, as outlined in the protocol.
* All participants must have measurable diseases per central laboratory as outlined in protocol

Exclusion Criteria:

* Has received prior etentamig treatment.
* Prior exposure to BCMA-targeted therapy as noted in the protocol.
* Has received prior cereblon E3 ligase modulatory drug (CELMoD) (iberdomide or mezigdomide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2036-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose-Limiting Toxicities (DLT)s of Etentamig when given in Combination with Iberdomide in Participants with Relapsed/Refractory Multiple Myeloma (RRMM) | Up to Approximately 56 Days
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Number of Participants with Adverse Events (AE)s | Up to Approximately 129 Months
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Partial Response (PR) Response Rate (RR) | Up to 3 Years
  PR is defined >= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hours, if the serum and urine M-protein are unmeasurable, a >= 50% decrease in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, if the serum and urine M-protein are unmeasurable, and serum free light assay is also unmeasurable, a >= 50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >= 30%, >= 50% reduction in the size of soft tissue plasmacytomas is also required, if present at baseline.
Very Good Partial Response (VGPR) RR | Up to 3 Years
  VGPR is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or >= 90% reduction in serum M-protein plus urine M-protein < 100 mg per 24 hours, for participants in whom the only measurable disease is by serum free light chains (FLC) levels, VGPR is defined as >= 90% decrease in the difference between involved and uninvolved FLC levels.
Complete Response (CR) RR | Up to 3 Years
  CR is defined negative immunofixation on the serum and urine (regardless of whether disease at baseline was measurable on serum, urine, both, or neither), disappearance of any soft tissue plasmacytomas, < 5% plasma cells in bone marrow, and for participants in whom the only measurable disease is by serum FLC levels, a normal FLC ratio is also required.
Stringent Complete Response (sCR) RR | Up to 3 Years
  sCR is defined negative immunofixation on the serum and urine (regardless of whether disease at baseline was measurable on serum, urine, both, or neither), disappearance of any soft tissue plasmacytomas, < 5% plasma cells in bone marrow, normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry (kappa/lambda ratio <= 4:1 or >= 1:2 for kappa and lambda participants, respectively, after counting >= 100 plasma cells).
Overall Response Rate (ORR) | Up to 3 Years
  ORR (PR + VGPR + CR + sCR) will be defined as the proportion of participants who achieved a PR or better.
Progression-Free Survival (PFS) | Up to 3 Years
  PFS is defined as the number of days from the date of first dose to the date of earliest disease progression or death.
Duration of Response (DOR) | Up to 3 Years
  DOR is defined as the number of days from the date of first response (sCR, CR, VGPR, or PR) to the earliest recurrence, progressive disease, or death, whatever occurs first.
Time-to-Progression (TTP) | Up to 3 Years
  TTP will be defined as the number of days from the date of first dose to the date of earliest disease progression.
Minimal Residual Disease (MRD) negativity | Up to 3 Years
  The MRD negativity rate is defined as the proportion of participants who achieve MRD negative status.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (7):
  - Beverly Hills Cancer Center /ID# 266921, Beverly Hills, California
  - Colorado Blood Cancer Institute /ID# 273751, Denver, Colorado
  - Washington University /ID# 266972, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey /ID# 266833, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center - New York - York Avenue /ID# 270282, New York, New York
  - University Of North Carolina Health Care - Hillsborough Campus /ID# 278230, Hillsborough, North Carolina
  - Swedish Cancer Institute /ID# 268052, Seattle, Washington
- Australia (5):
  - Blacktown Hospital /ID# 265983, Blacktown, New South Wales
  - Wollongong Hospital /ID# 265625, Wollongong, New South Wales
  - The Alfred Hospital /ID# 265981, Melbourne, Victoria
  - Austin Hospital /ID# 265984, Melbourne, Victoria
  - Sir Charles Gairdner Hospital /ID# 265985, Nedlands, Western Australia
- Canada (2):
  - University Health Network_Princess Margaret Cancer Centre /ID# 275636, Toronto, Ontario
  - Jewish General Hospital /ID# 267574, Montreal, Quebec
- France (5):
  - Chu de Nice-Hopital Larchet Ii /Id# 266845, Nice, Alpes-Maritimes
  - Hôpital La Timone /ID# 267053, Marseille, Bouches-du-Rhone
  - Chu De Lille - Hopital Claude Huriez /ID# 270193, Lille, Hauts-de-France
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau /ID# 267694, Tours, Indre-et-Loire
  - IUCT Oncopole /ID# 266391, Toulouse, Occitanie
- Japan (4):
  - Kumamoto University Hospital /ID# 270530, Kumamoto, Kumamoto
  - Dokkyo Medical University Hospital /ID# 271648, Mibu, Tochigi
  - Nippon Medical School Hospital /ID# 270254, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 268342, Koto-ku, Tokyo
- Netherlands (2):
  - Amsterdam UMC, Location VUmc /ID# 267670, Amsterdam, North Holland
  - Universitair Medisch Centrum Utrecht /ID# 267660, Utrecht
- Oslo Universitetssykehus Ulleval /ID# 275433, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-555